CLINICAL TRIAL: NCT00072553
Title: A Phase II Of An Optimized LV-5FU-Oxaliplatin Strategy With Celebrex In Metastatic Colorectal Cancer, Optimox2-Celecoxib Study
Brief Title: Celecoxib, Leucovorin, Fluorouracil, and Oxaliplatin in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000340181; GERCOR-OPTIMOX2-CELECOXIB-2002; EU-20325
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
Keywords: stage IV rectal cancer; stage IV colon cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent rectal cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — Celecoxib; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: celecoxib
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as leucovorin, fluorouracil, and oxaliplatin, use different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of colorectal cancer by stopping blood flow to the tumor and by blocking the enzymes necessary for tumor cell growth. Combining chemotherapy with celecoxib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining celecoxib with leucovorin, fluorouracil, and oxaliplatin in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic colorectal cancer treated with celecoxib, leucovorin calcium, fluorouracil, and oxaliplatin.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the time of disease control to evaluate progression-free survival in patients treated with this regimen.
* Determine the salvage surgery rate in patients treated with this regimen.
* Determine the duration of chemotherapy-free intervals in patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive FOLFOX7 chemotherapy comprising oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. Patients also receive oral celecoxib twice daily beginning on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease stop treatment. If disease progression occurs during the chemotherapy-free interval, patients receive an additional 6 courses.

Patients with responding disease after receiving at least 6 courses of chemotherapy may undergo surgery. Beginning within 10 weeks after surgery, patients receive simplified LV5FU2 chemotherapy comprising leucovorin calcium IV over 2 hours on day 1, fluorouracil IV over 46 hours beginning on day 1, and oral celecoxib twice daily beginning on day 1. Treatment repeats every 14 days for at least 12 courses.

Quality of life is assessed at baseline, during courses 4 and 6, and then every 2 months thereafter.

Patients are followed at 1 month and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Metastatic disease
  * Inoperable disease (i.e., not suitable for complete carcinological surgical resection)
* Measurable disease or nonmeasurable disease

  * At least 1 unidimensionally measurable lesion at least 20 mm by conventional CT scan OR 10 mm by spiral CT scan
  * Nonmeasurable disease defined as all other lesions, including small lesions or truly nonmeasurable disease
* No CNS metastases
* No exclusive bone metastases
* No symptomatic ascites or pleural effusion not evacuated before study entry

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No known significant bleeding disorder

Hepatic

* Alkaline phosphatase less than 3 times upper limit of normal (ULN)

Renal

* Creatinine less than 1.5 times ULN OR
* Creatinine clearance at least 30 mL/min
* No uncontrolled hypercalcemia

Cardiovascular

* No congestive heart failure

Gastrointestinal

* No total or partial bowel obstruction
* No active gastric or duodenal ulceration or gastrointestinal bleeding within the past year
* No active inflammatory bowel disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No peripheral sensory neuropathy
* No known sensitivity to celecoxib, other COX-2 inhibitors, NSAIDs, salicylates, or sulfonamides
* No AIDS-related illness
* No active infection
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for metastatic disease

Chemotherapy

* Prior adjuvant chemotherapy allowed provided the progression-free interval after completion of therapy is more than 6 months in duration
* No prior chemotherapy for metastatic disease
* No prior adjuvant oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent chronic oral or IV corticosteroid use (i.e., 2 weeks or longer in duration)

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational drugs
* No other concurrent investigational drugs or treatments
* No concurrent prophylactic fluconazole
* No concurrent chronic full-dose aspirin (at least 325 mg/day), other nonsteroidal anti-inflammatory drugs (NSAIDs), or other cyclooxygenase (COX)-2 inhibitors

  * Concurrent low-dose (cardioprotective) aspirin (80 mg/day or equivalent) allowed
* No concurrent lithium
* No other concurrent anticancer therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Toxicity
Time of disease control (progression-free survival)
Salvage surgery rate
Duration of chemotherapy-free intervals
Tolerability
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Andre, MD, Study Chair — GERCOR - Multidisciplinary Oncology Cooperative Group
Locations (1):
- Hopital Tenon, Paris, France

REFERENCES:
- [Result] Andre T, Tournigand C, Mineur L, Fellague-Chebra R, Flesch M, Mabro M, Hebbar M, Postel Vinay S, Bidard FC, Louvet C, de Gramont A. Phase II study of an optimized 5-fluorouracil-oxaliplatin strategy (OPTIMOX2) with celecoxib in metastatic colorectal cancer: a GERCOR study. Ann Oncol. 2007 Jan;18(1):77-81. doi: 10.1093/annonc/mdl336. Epub 2006 Oct 9. PMID 17030548